CLINICAL TRIAL: NCT06170645
Title: Transcutaneous Vagus Nerve Stimulation as a Complementary Therapy to Exercise in Chronic Fatigue: Single-center, Controlled, Randomized, Blinded Study
Brief Title: Transcutaneous Vagus Nerve Stimulation as a Complementary Therapy to Exercise in Chronic Fatigue
Acronym: PAF-tVNS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 23CH153; 2023-A01792-43 (Other: ANSM)
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Chronic Fatigue Syndrome
Keywords: Chronic fatigue; Transcutaneous vagal nerve stimulation (tVNS); adapted physical activity (APA)
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with active tVNS (Experimental): Patients consulting on St Etienne hospital and suffering from fibromyalgia and long Covid will be included.
  Interventions: Other: APA program; Other: Active transcutaneous VNS
- Patients with sham tVNS (Sham Comparator): Patients consulting on St Etienne hospital and suffering from fibromyalgia and long Covid will be included.
  Interventions: Other: APA program; Other: Sham transcutaneous VNS

INTERVENTIONS:
Other: APA program — An APA program of 12 weeks, 2 sessions of 1h/week for mixed endurance, strengthening and stretching work. The program can be realized at home or in structure.
Other: Active transcutaneous VNS — After each APA session, a 1h-tVNS session is delivered on the conchae aurea of the left ear, in resting condition. Parameters of tVNS : frequency 20Hz, impulsion 200ms, amplitude 1mA below the unpleasant sensation level.
  Arms: Patients with active tVNS
Other: Sham transcutaneous VNS — After each APA session, a 1h-tVNS session is delivered on the left earlobe, in resting condition. Parameters of tVNS : frequency 20Hz, impulsion 200ms, amplitude 1mA below the unpleasant sensation level.
  Arms: Patients with sham tVNS

SUMMARY:
Chronic fatigue is enhanced by adapted physical activity (APA) programs. Patients consulting on St Etienne hospital and suffering from fibromyalgia and long Covid benefit from a 4-6 week APA program, with 2 sessions per week. While most patients are improved by these exercise-training programs, for some the benefits remain very modest, and patients describe persistent fatigue. The literature unanimously describes the necessity of longer APA protocols (8-12 weeks, 2-3 sessions/week) for fatigue reduction in fibromyalgia and long Covid. However, it seems difficult to adhere to an optimal program as described in the literature for these fatigued patients. The investigators want to test a device that would both reduce fatigue and improve recovery between APA sessions, in order to gradually reach the recommendations for APA practice. Transcutaneous vagal nerve stimulation (tVNS) seems to be a promising approach. Thus, combining an APA intervention with a tVNS protocol could potentiate the expected and now well-known effect of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Signature of informed consent
* Confirmed diagnosis of fibromyalgia or long Covid (ACR 2016 criteria and persistent symptoms lasting more than 6 months after a positive RT-PCR test, respectively)
* Persistent fatigue after an exercise rehabilitation program (FSS score > 36)
* Physical inactivity, i.e. <150 minutes per week of physical activity

Exclusion Criteria:

* Pre-existing atrial fibrillation,
* Left ventricular ejection fraction <40%
* Severe heart failure
* Recent stroke or myocardial infarction (<6 months)
* Unilateral or bilateral vagotomy
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Fatigue evaluation assessed by autonomic nervous system activity | Month : 0; 3
  The root mean square of successive differences in heart rate (in milliseconds) will be measured from a nocturnal Holter ECG recording (Novacor, Paris, France) at the end of the 3-month APA and tVNS programme (month 3) and compared with pre-programme values (inclusion).

SECONDARY OUTCOMES:
Fatigue Severity Scale (FSS) | Month : 0; 6
  Subjective fatigue assessed by FSS, score from 9 to 63. The higher the score, the more severe the fatigue is and the more it affects the person's activities.
Medical Outcome Study Short Form questionnaire (MOS-SF 12) | Month : 0; 6
  Quality of life assessed by the MOS-SF 12 questionnaire , score from 0 to 100. A low score reflects a perception of poor health, loss of function and the presence of pain. A high score reflects a perception of good health, absence of functional deficit and pain.
Pittsburgh questionnaire | Month : 0; 6
  Quality of sleep assessed by Pittsburgh questionnaire (score 0 to 21). The 7 components of the score add up to give an overall score ranging from give an overall score ranging from 0 to 21 points, with 0 meaning that there are no difficulties, and 21 indicating major difficulties.
6-minute walk test (6MWT) | Month : 0; 6
  Physical condition assessed by the walking distance covered in the 6MWT, walking distance in m.
Adult Physical Activity Questionnaire (APAQ) | Month : 0; 6
  Physical activity assessed by the APAQ, time spend to physical activity in hours/day.
Step count per day | Month : 0; 6
  Objective physical activity assessed by step count per day using a Garmin Vivofit 4 activity tracker.
Ratio of Low Frequency to High Frequency (LF/HF) | Month : 0; 6
  The autonomic balance (sympathetic/parasympathetic) will be analysed by measuring the LF/HF ratio on the basis of a nocturnal Holter ECG recording (Novacor, Paris, France).

CONTACTS AND LOCATIONS:
Overall Officials: David HUPIN, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Centre Hospitalier de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No